CLINICAL TRIAL: NCT01793766
Title: Neurobehavioral Contribution to Weight Loss Maintenance: an Interdisciplinary Experimental Study With Noninvasive Brain Modulation
Brief Title: Non-invasive Brain Modulation for Weight Maintenance
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Nutrition and Obesity Research Center at Harvard (NORC-H) (Unknown)
Responsible Party: Principal Investigator, Takara Stanley, M.D., Assistant Professor of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2013-P-000191
Record Dates: First submitted 2013-02-08; First posted 2013-02-18 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brain modulation (Experimental): 10 sessions of brain modulation with Eldith/Neuroconn transcranial Direct Current Stimulation device
  Interventions: Device: Brain modulation
- Placebo (sham modulation) (Placebo Comparator): 10 placebo sessions where no brain modulation takes place
  Interventions: Device: Sham modulation

INTERVENTIONS:
Device: Brain modulation — Brain modulation using Eldith/Neuroconn transcranial Direct Current Stimulation device
  Arms: Brain modulation
Device: Sham modulation
  Arms: Placebo (sham modulation)

SUMMARY:
This is a study of overweight men and women. Everybody will receive a very low calorie diet to eat in place of meals for 10 weeks. During the last two weeks of the diet, half of the patients will receive an intervention to activate parts of their brain that can help them eat less. The other half of the patient will receive a placebo or sham intervention. The intervention will involve a small electric current given every day for 10 days. Everybody will be monitored for 16 more weeks (total of 26 weeks) while on a weight maintenance diet to see if the intervention helps people keep the weight off.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 20-55 years old
2. BMI 30-50 kg/m2
3. Willing to undergo 10 week supervised VLCD

Exclusion Criteria:

1. Obesity due to a known secondary cause (Cushing's syndrome, hypothyroidism, etc) or a history of weight loss surgery
2. Subjects who have a known history of diabetes, fasting blood sugar >125 mg/dl or using any anti-diabetic drugs
3. Changes in lipid lowering or anti-hypertensive regimen within 3 months of screening
4. Hemoglobin <10 g/dL, Creatinine >1.5 mg/dL
5. QT interval >440 ms on EKG
6. Subjects with unstable psychiatric conditions as assessed by a psychologist
7. Allergy or intolerance to components of the mixed meal challenge
8. Additional contraindications to receive transcranial direct current stimulation (tDCS):

   1. Personal or family history of seizures, epilepsy or other unexplained loss of consciousness.
   2. Current or past history of skin disease or damaged skin on the scalp at the site of stimulation (i.e. eczema, skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc.).
   3. Prior neurosurgical procedure or radiation treatment to the brain.
   4. Known diagnosis of brain lesions, such as tumor, stroke or multiple sclerosis
   5. Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, ventriculoperitoneal shunt or any metallic implant on the head.

   (Note: Intake of centrally acting medications will be allowed, as there is no evidence that any medication can increase the risk of adverse effects during tDCS.)
9. Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit
10. Any condition judged by the patient's physician to cause this clinical trial to be detrimental to the patient

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in weight from week 11 to 26 | Week 11 to 26
  Patients will be placed on a very low calorie diet from baseline to week 11. The primary end point is the maintenance of weight loss from week 11 to week 26 after the very low calorie diet is stopped.

SECONDARY OUTCOMES:
Change in appetite hormones on mixed meal challenge test | Week 0 to 8, 11 and 26
  Appetite hormones such as ghrelin change in response to nutrition. Dieting increases ghrelin and decreases other appetite hormones. We will assess if the brain modulation intervention will prevent the dieting induced increase in ghrelin and changes in other appetite hormones.
Change in appetite | Week 0 to 8, 11, 18 and 26
  Degree of hunger (or satiety) can be assessed by use of visual analog scale and monitoring food intake diaries and questionnaires. We will assess if the brain modulation intervention can prevent the diet induced increases in appetite using the visual analog scale, food diary and questionnaires.
Change in body composition | Week 0 to 8 and 26
  Weight loss can affect both fat mass and muscle (lean) mass. We will assess if the weight loss by low-calorie diet and weight maintenane facilitated by brain modulation will preferentially affect fat mass or lean mass by use of dual energy X-ray absorptiometry.
Change in metabolic parameters | Week 0 to 8, 11, 18, 26
  Weight loss and successful weight loss maintenance can improve insulin resistance (risk for diabetes mellitus) and cholesterol profile. We will assess the changes in risk for diabetes and cholesterol from the low-calorie diet and brai modulation mediated weight maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Takara Stanley, MD, Principal Investigator — Massachusetts General Hospital; Miguel Alonso-Alonso, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Winfield S. Butsch, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No